CLINICAL TRIAL: NCT00811421
Title: Evaluation of the Safety and Efficacy of Mefloquine as Intermittent Preventive Treatment of Malaria in Pregnancy
Brief Title: Evaluation of Alternative Antimalarial Drugs for Malaria in Pregnancy
Acronym: MiPPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Barcelona Centre for International Health Research (Other); Institute of Tropical Medicine, University of Tuebingen (Other); Institut de Recherche pour le Developpement (Other Government); Université d'Abomey-Calavi (Other); Albert Schweitzer Hospital (Other); Kenya Medical Research Institute (Other); Ifakara Health Institute (Other); Centro de Investigacao em Saude de Manhica (Other); Vienna School of Clinical Research (VSCR), Austria. (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Malaria in Pregnancy Consortium (Other)
Responsible Party: Professor Clara Menendez Santos, Barcelona Centre for International Health Research (CRESIB), Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IP.07.31080.002
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Pregnancy; Malaria; HIV Infections
Keywords: Malaria; Pregnancy; HIV; Prevention; Malaria prevention
MeSH Terms: conditions — Malaria; HIV Infections | interventions — fanasil, pyrimethamine drug combination; Mefloquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Trial 1: IPTp-SP+LLITNs (Active Comparator): HIV-negative pregnant women receiving 2 doses of IPTp (500mg of sulfadoxine and 25 mg of pyrimethamine) in the context of long lasting Insecticide Treated Nets (LLITNs)
  Interventions: Drug: Sulphadoxine-pyrimethamine
- Trial 1: IPTp-MQ (full dose) + LLITNs (Experimental): HIV-negative pregnant women receiving 2 full doses of IPTp (15 mg/Kg) in the context of long lasting Insecticide Treated Nets (LLITNs)
  Interventions: Drug: Mefloquine (full dose)
- Trial 1: IPTp-MQ (split dose)+LLITNs (Experimental): HIV-negative pregnant women receiving 2 doses of MQ as IPTp split dose over 2 days (15mg/kg) in the context of long lasting Insecticide Treated Nets (LLITNs
  Interventions: Drug: Mefloquine (split dose)
- Trial 2: CTX+IPTp-Placebo+LLITNs (Experimental): HIV-positive pregnant women receiving 3 doses of IPTp (placebo) in the context of long lasting Insecticide Treated Nets (LLITNs)
  Interventions: Drug: placebo
- Trial 2: CTX + IPTp-MQ+ LLITNs (Experimental): HIV-positive pregnant women receiving 3 doses of IPTp (15 mg/Kg) in the context of long lasting Insecticide Treated Nets (LLITNs)
  Interventions: Drug: mefloquine

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine — SP oral administration (500mg sulphadoxine and 25mg pyrimethamine) as IPTp at the 1st and 2nd Antenatal Clinic visit
  Arms: Trial 1: IPTp-SP+LLITNs
Drug: Mefloquine (full dose) — MQ oral administration (15 mg/Kg) on 1 day at the 1st and 2nd Antenatal Clinic visit as IPTp
  Arms: Trial 1: IPTp-MQ (full dose) + LLITNs
Drug: Mefloquine (split dose) — MQ oral administration (15 mg/kg) split dose over 2 days at the 1st and 2nd ANC visit as IPTp
  Arms: Trial 1: IPTp-MQ (split dose)+LLITNs
Drug: placebo — MQ-placebo oral administration at the 1st, 2nd and 3rd Antenatal Clinic visit as IPTp
  Arms: Trial 2: CTX+IPTp-Placebo+LLITNs
Drug: mefloquine — MQ oral administration (15 mg/Kg) at the 1st and 2nd Antenatal Clinic visit as IPTp
  Arms: Trial 2: CTX + IPTp-MQ+ LLITNs

SUMMARY:
The study aims at comparing the safety, tolerability and efficacy of Mefloquine (MQ) to Sulfadoxine-Pyrimethamine (SP) as Interment Preventive Treatment in pregnancy (IPTp) for the prevention of malaria effects on the mother and her infant.

DETAILED DESCRIPTION:
The current recommendation by the World Health Organization (WHO) to prevent malaria infection in pregnancy in areas of stable malaria transmission relies on:

* Prompt and effective case management of malaria illness
* The use of intermittent preventive treatment (IPTp) with at least 2 treatment doses of sulfadoxine-pyrimethamine (SP) and
* The use of insecticide treated nets (ITNs)

However, the spread of parasite resistance to SP, particularly in eastern Africa, and the significant overlap in some regions of malaria transmission and high prevalence of HIV infection, have raised concerns about the medium and long-term use of SP for IPTp.

HIV infection increases susceptibility to malaria and may reduce the efficacy of interventions. The evaluation of alternative antimalarials for IPTp is thus urgently needed also involving HIV infected women.

Of all the current available alternative antimalarial drugs, mefloquine (MQ) is the one that offers the most comparative advantages to SP.

A randomized multicenter trial will be conducted in 4 sites in Africa (Benin, Gabon, Tanzania and Mozambique) in order to compare the safety and efficacy of SP versus MQ as IPTp in the context of ITNs. In addition, MQ tolerability will be also evaluated by comparing the administration of MQ as a single intake with its administration as split dose in two days. In total 4716 pregnant women will be enrolled at the antenatal clinic (ANC) and will be followed until the infant is one year old.

Besides, in those countries where HIV prevalence in pregnant women is > 10%, MQ-IPTp will be compared to Placebo-IPTp in HIV infected pregnant women receiving cotrimoxazole (CTX) prophylaxis. This trial will be double blinded and will be carried out in Kenya, Tanzania and Mozambique. It will involve 1070 pregnant women that will be followed until the infant is 2 months old.

ELIGIBILITY:
Inclusion Criteria:

Trial 1:

* Permanent resident in the area
* Gestational age at the first antenatal visit ≤ 28 weeks
* Signed informed consent
* Agreement to deliver in the study site's maternity(ies) wards

Trial 2:

* Permanent resident in the area.
* Gestational age at the first antenatal visit ≤ 28 weeks
* HIV seropositive (after voluntary counseling and testing)
* Indication to receive CTX prophylaxis (according to the national guidelines)
* Signed informed consent
* Agreement to deliver in the study site's maternity(ies) wards.

Exclusion Criteria:

Trial 1:

* Residence outside the study area or planning to move out in the following 18 months from enrollment
* Gestational age at the first antenatal visit > 28 weeks of pregnancy
* Known history of allergy to sulfa drugs or mefloquine
* Known history of severe renal, hepatic, psychiatric or neurological disease
* MQ or halofantrine treatment in the preceding 4 weeks
* HIV infection
* Participating in other studies

Trial 2:

* Residence outside the study area or planning to move out in the following 10 months from enrollment
* Gestational age at the first antenatal visit > 28 weeks of pregnancy
* Known history of allergy to CTX or MQ
* Known history of severe renal, hepatic, psychiatric or neurological disease
* MQ or halofantrine treatment in the preceding 4 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5820 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Trial 1 (IPTp MQ vs IPTp SP): Low birth weight. | day 0, birth
Trial 2 (CTX+IPTp MQ vs. CTX+IPTp placebo): Peripheral parasitaemia. | day 0, delivery

SECONDARY OUTCOMES:
Trial 1: Prevalence of placental P. falciparum infection. Prevalence of moderate maternal anaemia at delivery. | day 0, delivery
Trial 2: Prevalence of placental P. falciparum infection. Prevalence of low birth weight babies (< 2500 g). | day 0, birth

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Barcelona Centre for International Health Research
Locations (5):
- Faculté des Sciences de la Santé (FSS), Université d'Abomey Calavi, Allada, Benin
- Medical Rsearch Unit (MRU), Albert Schweitzer Hospital, Lambaréné, Gabon
- Kenya Medical Research Institute (KEMRI)/ CDC, Kisumu, Kenya
- Centro de Investigaçao em Saúde da Manhiça (CISM), Manhiça, Maputo Province, Mozambique
- Ifakara Health Institute (IHI), Dodoma, Tanzania

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Garrison A, Boivin MJ, Fievet N, Zoumenou R, Alao JM, Massougbodji A, Cot M, Bodeau-Livinec F. The Effects of Malaria in Pregnancy on Neurocognitive Development in Children at 1 and 6 Years of Age in Benin: A Prospective Mother-Child Cohort. Clin Infect Dis. 2022 Mar 9;74(5):766-775. doi: 10.1093/cid/ciab569. PMID 34297062
- [Derived] Zoleko-Manego R, Mischlinger J, Dejon-Agobe JC, Basra A, Mackanga JR, Akerey Diop D, Adegnika AA, Agnandji ST, Lell B, Kremsner PG, Matsiegui PB, Gonzalez R, Menendez C, Ramharter M, Mombo-Ngoma G. Birth weight, growth, nutritional status and mortality of infants from Lambarene and Fougamou in Gabon in their first year of life. PLoS One. 2021 Feb 9;16(2):e0246694. doi: 10.1371/journal.pone.0246694. eCollection 2021. PMID 33561169
- [Derived] Garrison A, Khoshnood B, Courtin D, Milet J, Garcia A, Massougbodji A, Ayotte P, Cot M, Bodeau-Livinec F. Blood lead level in infants and subsequent risk of malaria: A prospective cohort study in Benin, Sub-Saharan Africa. PLoS One. 2019 Jul 18;14(7):e0220023. doi: 10.1371/journal.pone.0220023. eCollection 2019. PMID 31318954
- [Derived] Mireku MO, Davidson LL, Zoumenou R, Massougbodji A, Cot M, Bodeau-Livinec F. Consequences of prenatal geophagy for maternal prenatal health, risk of childhood geophagy and child psychomotor development. Trop Med Int Health. 2018 Aug;23(8):841-849. doi: 10.1111/tmi.13088. Epub 2018 Jun 22. PMID 29876999
- [Derived] Moya-Alvarez V, Ouedraogo S, Accrombessi M, Cot M. High folate levels are not associated with increased malaria risk but with reduced anaemia rates in the context of high-dosed folate supplements and intermittent preventive treatment against malaria in pregnancy with sulphadoxine-pyrimethamine in Benin. Trop Med Int Health. 2018 Jun;23(6):582-588. doi: 10.1111/tmi.13064. Epub 2018 May 21. PMID 29683544
- [Derived] Ndam NT, Mbuba E, Gonzalez R, Cistero P, Kariuki S, Sevene E, Ruperez M, Fonseca AM, Vala A, Maculuve S, Jimenez A, Quinto L, Ouma P, Ramharter M, Aponte JJ, Nhacolo A, Massougbodji A, Briand V, Kremsner PG, Mombo-Ngoma G, Desai M, Macete E, Cot M, Menendez C, Mayor A. Resisting and tolerating P. falciparum in pregnancy under different malaria transmission intensities. BMC Med. 2017 Jul 17;15(1):130. doi: 10.1186/s12916-017-0893-6. PMID 28712360
- [Derived] Gonzalez R, Ruperez M, Sevene E, Vala A, Maculuve S, Bulo H, Nhacolo A, Mayor A, Aponte JJ, Macete E, Menendez C. Effects of HIV infection on maternal and neonatal health in southern Mozambique: A prospective cohort study after a decade of antiretroviral drugs roll out. PLoS One. 2017 Jun 2;12(6):e0178134. doi: 10.1371/journal.pone.0178134. eCollection 2017. PMID 28575010
- [Derived] Mireku MO, Davidson LL, Boivin MJ, Zoumenou R, Massougbodji A, Cot M, Bodeau-Livinec F. Prenatal Iron Deficiency, Neonatal Ferritin, and Infant Cognitive Function. Pediatrics. 2016 Dec;138(6):e20161319. doi: 10.1542/peds.2016-1319. Epub 2016 Nov 17. PMID 27940685
- [Derived] Mombo-Ngoma G, Mackanga JR, Gonzalez R, Ouedraogo S, Kakolwa MA, Manego RZ, Basra A, Ruperez M, Cot M, Kabanywany AM, Matsiegui PB, Agnandji ST, Vala A, Massougbodji A, Abdulla S, Adegnika AA, Sevene E, Macete E, Yazdanbakhsh M, Kremsner PG, Aponte JJ, Menendez C, Ramharter M. Young adolescent girls are at high risk for adverse pregnancy outcomes in sub-Saharan Africa: an observational multicountry study. BMJ Open. 2016 Jun 29;6(6):e011783. doi: 10.1136/bmjopen-2016-011783. PMID 27357200
- [Derived] Bodeau-Livinec F, Glorennec P, Cot M, Dumas P, Durand S, Massougbodji A, Ayotte P, Le Bot B. Elevated Blood Lead Levels in Infants and Mothers in Benin and Potential Sources of Exposure. Int J Environ Res Public Health. 2016 Mar 11;13(3):316. doi: 10.3390/ijerph13030316. PMID 26978384
- [Derived] Ruperez M, Gonzalez R, Mombo-Ngoma G, Kabanywanyi AM, Sevene E, Ouedraogo S, Kakolwa MA, Vala A, Accrombessi M, Briand V, Aponte JJ, Manego Zoleko R, Adegnika AA, Cot M, Kremsner PG, Massougbodji A, Abdulla S, Ramharter M, Macete E, Menendez C. Mortality, Morbidity, and Developmental Outcomes in Infants Born to Women Who Received Either Mefloquine or Sulfadoxine-Pyrimethamine as Intermittent Preventive Treatment of Malaria in Pregnancy: A Cohort Study. PLoS Med. 2016 Feb 23;13(2):e1001964. doi: 10.1371/journal.pmed.1001964. eCollection 2016 Feb. PMID 26905278
- [Derived] Mireku MO, Davidson LL, Koura GK, Ouedraogo S, Boivin MJ, Xiong X, Accrombessi MM, Massougbodji A, Cot M, Bodeau-Livinec F. Prenatal Hemoglobin Levels and Early Cognitive and Motor Functions of One-Year-Old Children. Pediatrics. 2015 Jul;136(1):e76-83. doi: 10.1542/peds.2015-0491. Epub 2015 Jun 8. PMID 26055847
- [Derived] Sicuri E, Fernandes S, Macete E, Gonzalez R, Mombo-Ngoma G, Massougbodgi A, Abdulla S, Kuwawenaruwa A, Katana A, Desai M, Cot M, Ramharter M, Kremsner P, Slustker L, Aponte J, Hanson K, Menendez C. Economic evaluation of an alternative drug to sulfadoxine-pyrimethamine as intermittent preventive treatment of malaria in pregnancy. PLoS One. 2015 Apr 27;10(4):e0125072. doi: 10.1371/journal.pone.0125072. eCollection 2015. PMID 25915616
- [Derived] Gonzalez R, Desai M, Macete E, Ouma P, Kakolwa MA, Abdulla S, Aponte JJ, Bulo H, Kabanywanyi AM, Katana A, Maculuve S, Mayor A, Nhacolo A, Otieno K, Pahlavan G, Ruperez M, Sevene E, Slutsker L, Vala A, Williamsom J, Menendez C. Intermittent preventive treatment of malaria in pregnancy with mefloquine in HIV-infected women receiving cotrimoxazole prophylaxis: a multicenter randomized placebo-controlled trial. PLoS Med. 2014 Sep 23;11(9):e1001735. doi: 10.1371/journal.pmed.1001735. eCollection 2014 Sep. PMID 25247995
- [Derived] Gonzalez R, Mombo-Ngoma G, Ouedraogo S, Kakolwa MA, Abdulla S, Accrombessi M, Aponte JJ, Akerey-Diop D, Basra A, Briand V, Capan M, Cot M, Kabanywanyi AM, Kleine C, Kremsner PG, Macete E, Mackanga JR, Massougbodgi A, Mayor A, Nhacolo A, Pahlavan G, Ramharter M, Ruperez M, Sevene E, Vala A, Zoleko-Manego R, Menendez C. Intermittent preventive treatment of malaria in pregnancy with mefloquine in HIV-negative women: a multicentre randomized controlled trial. PLoS Med. 2014 Sep 23;11(9):e1001733. doi: 10.1371/journal.pmed.1001733. eCollection 2014 Sep. PMID 25247709